CLINICAL TRIAL: NCT00687687
Title: A Phase II Evaluation of Paclitaxel (Taxol, NSC #673089), Carboplatin (Paraplatin, NSC #241240), and BSI-201 (NSC #746045, IND #71,677) in the Treatment of Advanced, Persistent, or Recurrent Uterine Carcinosarcoma
Brief Title: Evaluation of Paclitaxel (Taxol, NSC #673089), Carboplatin (Paraplatin, NSC #241240), and BSI-201 (NSC #746045, IND #71,677) in the Treatment of Advanced, Persistent, or Recurrent Uterine Carcinosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Gynecologic Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCD11615; GOG 0232C; 20070103 (Other: BiPar); NCT00588744 (obsolete NCT alias)
Expanded Access: NCT01130259 (No longer available)
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Uterine Carcinosarcoma
Keywords: Patients must have advanced (stage III or IV), persistent or recurrent uterine carcinosarcoma with documented disease progression.
MeSH Terms: interventions — Paclitaxel; Carboplatin; iniparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pacitaxel/Carboplatin/Iniparib (Experimental): Participants will be administered pacitaxel, carboplatin and BSI-201 (Iniparib) in 21 day treatment cycles. Treatment will continue until disease progression or adverse effects prohibit further therapy.
  Interventions: Drug: paclitaxel; Drug: carboplatin; Drug: BSI-201 (Iniparib)

INTERVENTIONS:
Drug: paclitaxel — Paclitaxel will be administered IV over 3 hours on Day 1 every 21 days.
Drug: carboplatin — Carboplatin will be administered intravenously (IV) over 30 minutes on day 1 after pacitaxel administration, every 21 days.
Drug: BSI-201 (Iniparib) — BSI-201 will be administered IV over one hour twice weekly beginning on day 1 (doses of BSI-201 must be separated by at least 2 days).
  Other Names: SAR204550

SUMMARY:
To estimate the antitumor activity of paclitaxel, carboplatin, plus BSI-201 in patients with recurrent or advanced uterine carcinosarcomas.

Based on data generated by BiPar/Sanofi, it is concluded that iniparib does not possess characteristics typical of the PARP inhibitor class. The exact mechanism has not yet been fully elucidated, however based on experiments on tumor cells performed in the laboratory, iniparib is a novel investigational anti-cancer agent that induces gamma-H2AX (a marker of DNA damage) in tumor cell lines, induces cell cycle arrest in the G2/M phase in tumor cell lines, and potentiates the cell cycle effects of DNA damaging modalities in tumor cell lines. Investigations into potential targets of iniparib and its metabolites are ongoing.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have advanced (stage III or IV), persistent or recurrent uterine carcinosarcoma with documented disease progression. Histologic confirmation of the original primary tumor is required.
* All patients must have measurable disease. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest dimension to be recorded). Each lesion must be greater than 20 mm when measured by conventional techniques, including palpation, plain x-ray, CT, and MRI, or greater than 10 mm when measured by spiral CT.
* Patients must have at least one "target lesion" to be used to assess response on this protocol as defined by RECIST (Section 8.1). Tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy.
* Patients must have a GOG Performance Status of 0, 1, or 2.
* Adequate bone marrow,renal, hepatic, and neurological function

Exclusion Criteria:

* Patients who have received prior cytotoxic chemotherapy for management of uterine carcinosarcoma.
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer and other specific malignancies as noted in Sections 3.23 and 3.24 are excluded if there is any evidence of other malignancy being present within the last five years. Patients are also excluded if their previous cancer treatment contraindicates this protocol therapy.
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis OTHER THAN for the treatment of uterine carcinosarcoma within the last five years are excluded. Prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease.
* Patients MAY have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease.
* Patients who have symptomatic or untreated brain metastases requiring concurrent treatment, inclusive of but not limited to surgery, radiation, and corticosteroids.
* Patients who have a significant history of cardiac disease, i.e., myocardial infarction (MI) within 6 months of study registration, unstable angina, congestive heart failure (CHF) with New York Heart Association (NYHA) > class II, or uncontrolled hypertension.
* Patients who have a history of seizure disorder or are currently on anti-seizure medication.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-05; Primary Completion 2010-03 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Clinical response rate | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (37):
- United States (37):
  - Research Site, Aurora, Colorado
  - Research Site, Englewood, Colorado
  - Research Site, New Britain, Connecticut
  - Research Site, Orlando, Florida
  - Research Site, Gainsville, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Hinsdale, Illinois
  - Research Site, Urbana, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Scarborough, Maine
  - Research Site, Kalamazoo, Michigan
  - Research Site, Springfield, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Camden, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, Buffalo, New York
  - Research Site, New York, New York
  - Research Site, Stony Brook, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Mentor, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Abington, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Wynnewood, Pennsylvania
  - Research Site, Wyomissing, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Burlington, Vermont
  - Research Site, Richmond, Virginia
  - Research Site, Roanoke, Virginia
  - Research Site, Madison, Wisconsin

REFERENCES:
- [Derived] Aghajanian C, Sill MW, Secord AA, Powell MA, Steinhoff M. Iniparib plus paclitaxel and carboplatin as initial treatment of advanced or recurrent uterine carcinosarcoma: a Gynecologic Oncology Group Study. Gynecol Oncol. 2012 Sep;126(3):424-7. doi: 10.1016/j.ygyno.2012.05.024. Epub 2012 May 24. PMID 22634397